CLINICAL TRIAL: NCT03014687
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Study Evaluating the Impact of Prophylactic Oral Antibiotics on Sinonasal Outcomes Following Endoscopic Transsphenoidal Surgery for Pituitary Lesions
Brief Title: Prophylactic Oral Antibiotics on Sinonasal Outcomes Following Endoscopic Transsphenoidal Surgery for Pituitary Lesions
Acronym: POET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Thomas Jefferson University (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Pam Dewey, Research Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHX-16-0134-30-12
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Antibiotics; Pituitary Adenoma
Keywords: transsphenoidal surgery
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Trimethoprim; Sulfamethoxazole; Cefdinir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Nasal Care (Placebo Comparator): One dose of preoperative intravenous (iv) antibiotic (e.g., cefazolin 1gm, or cefuroxime 1.5gm, or clindamycin 300mg will be administered within 60 minutes of start of surgery. Repeat intraoperative dosing of antibiotics is permitted if length of surgery exceeds recommended dosing interval. IV antibiotic dosing schedules: Cefazolin 1 gm iv Q6 hr -or- Cefuroxime 1.5gm iv Q8 hr -or- Clindamycin 300 mg iv Q12 hr. Postoperative antibiotics: Study participants will receive one dose only of postoperative intravenous antibiotic (e.g., cefazolin 1gm, or cefuroxime 1.5gm, or clindamycin 300mg [cephalosporin allergic patients]) according to the recommended dosing schedule described above. This dose of antibiotics is in addition to the preoperative dose. Placebo PO BID (twice daily) will commence on the morning of postoperative day 1 and continue for 7 days.
  Interventions: Drug: Placebo
- Standard Nasal Care + Oral Antibiotics (Experimental): One dose of preoperative iv antibiotic (cefazolin 1gm, or cefuroxime 1.5gm, or clindamycin 300mg) will be administered within 60 minutes of start of surgery. Repeat intraoperative dosing of antibiotics is permitted if length of surgery exceeds recommended dosing interval. IV antibiotic dosing schedules: Cefazolin 1 gm iv Q6 hr -or- Cefuroxime 1.5gm iv Q8 hr -or- Clindamycin 300 mg iv Q12 hr. Participants will receive 1 dose only of postoperative iv antibiotic (cefazolin 1gm, or cefuroxime 1.5gm, or clindamycin 300mg [cephalosporin allergic patients]) according to the recommended dosing schedule described above. This dose of antibiotics is in addition to the preoperative dose. Oral antibiotics will commence on the morning of postoperative day 1; this group will receive oral antibiotics (cefdinir [Omnicef®] 300 mg PO BID or trimethoprim/sulfamethoxazole [Bactrim DS™] PO BID for cephalosporin intolerant patients) for 7 days.
  Interventions: Drug: Oral Antibiotics cefdinir or trimethoprim/sulfamethoxazole

INTERVENTIONS:
Drug: Placebo — PO BID placebo for 7 days. Postoperative days 1 through 7: patients will administer saline spray (e.g., Ocean nasal spray) to both nostrils four times daily. Postoperative days 8 through 30: patients will begin twice daily sinus irrigation rinse (e.g., Neti-pot) until day 30. After day 30, patients will perform sinus irrigation as needed. If a patient is unable to tolerate nasal rinses, saline spray can be used as an alternative.
  Other Names: inert substance
  Arms: Standard Nasal Care
Drug: Oral Antibiotics cefdinir or trimethoprim/sulfamethoxazole — Oral antibiotics (cefdinir [Omnicef®] 300 mg PO BID or trimethoprim/sulfamethoxazole [Bactrim DS™] PO BID for cephalosporin intolerant patients) for 7 days.Postoperative days 1 through 7: patients will administer saline spray (e.g., Ocean nasal spray) to both nostrils four times daily. Postoperative days 8 through 30: patients will begin twice daily sinus irrigation rinse (e.g., Neti-pot) until day 30. After day 30, patients will perform sinus irrigation as needed. If a patient is unable to tolerate nasal rinses, saline spray can be used as an alternative.
  Other Names: Omnicef; Bactrim DS™ cephalosporin intolerant patients
  Arms: Standard Nasal Care + Oral Antibiotics

SUMMARY:
To find out whether oral antibiotics given after transsphenoidal endoscopic surgery for pituitary adenoma improves sinus and nasal symptoms, reduces the incidence of infection (sinusitis), and helps mucosal healing in the nasal passages.

DETAILED DESCRIPTION:
Transsphenoidal surgery is the standard of care for most symptomatic pituitary adenomas. Since transsphenoidal surgery exploits the nasal passage to reach the sella turcica and pituitary gland, the technique causes disruption of sinonasal function and temporarily impacts sinonasal quality of life. Disrupted sinonasal function is a primary source of postoperative morbidity following transsphenoidal surgery. Common sinonasal complications include sinusitis, synechiae formation, nasal obstruction and crusting. The development of postoperative sinusitis is specifically associated with decreased sinonasal function after surgery. Because the nasal cavity is a contaminated surgical field, practitioners routinely prescribe a course of oral postoperative antibiotics for 7-14 days (in addition to standard prophylactic perioperative intravenous antibiotics) with the intention of improving nasal functional outcomes. To date, no studies have examined whether the administration of oral antibiotics following transsphenoidal surgery improves sinonasal healing. This question has been studied in a closely-related field, functional endoscopic sinus surgery (FESS). A meta-analysis of clinical trial data obtained in FESS indicated that current literature does not support the use of oral antibiotics to reduce infection, improve symptoms scores, or improve endoscopic findings. Furthermore, there is the potential for antibiotic-related adverse events including the emergence of bacterial resistance, Clostridium difficile infection, and allergic reactions to the medication. Despite the lack of supporting evidence in FESS, prophylactic antibiotic use for improving sinonasal healing is still common in pituitary surgery. The investigators propose to study whether prophylactic oral antibiotics following transsphenoidal surgery improve sinonasal quality of life, reduce sinusitis incidence, and promote mucosal healing following endoscopic transsphenoidal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing endoscopic surgery for resection of pituitary tumors for nonfunctioning adenoma, acromegaly, or prolactinoma
* Adults >18 and <85 years of age
* English speaking and able to understand the ASK Nasal-12 and SNOT-22 scales
* Free of any physical, mental, or medical condition which, in the opinion of the investigator, makes study participation inadvisable

Exclusion Criteria:

* Anaphylaxis/intolerance to the study drugs
* Cirrhosis, hepatitis
* Any solid organ transplant or bone marrow transplant. And any patient felt to be immunocompromised by the investigators
* Renal failure on dialysis
* Any subject who is unwilling or unable to sign informed consent for the study
* Pregnancy
* Incarcerated patients
* Cushing's disease
* Rathke's Cleft cyst or pituitary cyst
* History of chronic sinusitis
* Anticipated use of nasal splints
* Anticipated use of nasal septal flap
* Active sinusitis
* Nasal polyps
* Previous sinus surgery
* Concurrent antibiotics for another indication (i.e., urinary tract infection)
* Immunodeficiency

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life from baseline - Anterior Skull Base Nasal Inventory 12 (ASK Nasal-12) | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Completed by subject in clinic or by phone interview. Assesses urge to blow nose; post-nasal discharge; thick nasal discharge; headaches; nose makes whistling sound; nasal crusting; trouble breathing through nose during day; trouble breathing through nose during night; not breathing equally in both nostrils; sense of smell; sense of taste; and, overall functioning of nose.Rating choices include no problem 0; very minor problem 1; minor problem 2; moderate problem 3; moderately severe problem 4; and, severe problem 5. Subject also selects the 5 symptoms/items listed that impact life the most.
Change in quality of life from baseline - Sino-Nasal Outcome Test (SNOT-22) | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Completed by subject in clinic or by phone interview. Assesses need to blow nose; nasal blockage; sneezing; runny nose; cough; post-nasal discharge; thick nasal discharge; ear fullness; dizziness; ear pain; facial pain/pressure; decreased sense of smell/taste; difficulty falling asleep; waking up at night; lack of a good night's sleep; wake up tired; fatigue; reduced productivity; reduced concentration; frustrated/restless/irritable; sad; and, embarrassed. Rating choices include no problem 0; very mild problem 1; mild or slight problem 2; moderate problem 3; severe problem 4; problem as bad as it can be 5. Subject also selects the 5 symptoms/items listed that impact life the most.

SECONDARY OUTCOMES:
Incidence of Acute Bacterial Sinusitis | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Incidence includes 3 or more of: i. Nasal congestion by patient report or physical exam, ii. Purulent nasal discharge by patient report or physical exam, iii. Facial pressure or pain or headache by patient report, iv. Antibiotics prescribed by a provider for the purpose of treating sinusitis.
Changes in endoscopic appearances using Postoperative Debridement Scoring Sheet (modified Lund-Kennedy score) | 1-2 and 3-4 weeks post-surgery
  Postoperative nasal endoscopy findings graded by surgeon. Grading includes Polyps = none 0; middle meatus 1; beyond middle meatus 2. Discharge = none 0; clear and thin 1; thick and purulent 2. Edema = none 0; mild 1; moderate 2; severe 3. Scarring = none 0; mild 1; moderate 2; severe 3. Crusting = none 0; mild 1; moderate 2; severe 3.
Sinusitis and antibiotic resistance as evidenced by nasal congestion | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Cultures and sensitivities when nasal congestion noted by patient report or physical exam.
Sinusitis and antibiotic resistance as evidenced by purulent discharge | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Cultures and sensitivities when purulent nasal discharge noted by patient report or physical exam.
Sinusitis and antibiotic resistance as evidenced by pressure | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Cultures and sensitivities when facial pressure noted by patient report.
Sinusitis and antibiotic resistance as evidenced by pain | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Cultures and sensitivities when facial pain noted by patient report.
Sinusitis and antibiotic resistance as evidenced headache | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, and 12 weeks post-surgery
  Cultures and sensitivities when headache noted by patient report.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Little, MD, Study Chair — Barrow Brain and Spine; James Evans, MD, Study Chair — Thomas Jefferson University
Locations (1):
- Barrow Brain and Spine, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided